CLINICAL TRIAL: NCT04584528
Title: Improving SCD Care Using Web-based Guidelines, Nurse Care Managers and Peer Mentors in Primary Care and Emergency Departments in Central North Carolina
Brief Title: Implementing an Individualized Pain Plan (IPP) for ED Treatment of VOE's in Sickle Cell Disease
Acronym: ALIGN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); RTI International (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Pro00073506_1; 5U01HL133964-05 (NIH)
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Sickle Cell Disease; Genetic Disease; Hematologic Diseases; Anemia, Sickle Cell
Keywords: sickle cell disease; vaso occlusive-episodes; Individualized Pain Plans; implementation science
MeSH Terms: conditions — Anemia, Sickle Cell; Genetic Diseases, Inborn; Hematologic Diseases | interventions — Electronic Health Records

STUDY DESIGN:
Intervention Model Description: Multi-site pre-post study design, with a core set of mandatory patient and provider intervention strategies for each participating site, and optional strategies to allow for intervention adaptation to local needs and resources.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EHR-embedded Individualized Pain Plan (IPP) (Other): The EHR embedded IPP will be made accessible to patients and ED providers at each study site.
  Interventions: Other: Electronic Health Record (EHR) Embedded Individualized Pain Plan (IPP)

INTERVENTIONS:
Other: Electronic Health Record (EHR) Embedded Individualized Pain Plan (IPP) — The IPPs will be developed by the Sickle Cell Disease providers at each study site based on patients' outpatient chronic opioid use and analgesic agent normally required for treatment of VOE in the ED. The Sickle Cell Disease provider will review the IPP with the patient, then upload the IPP to the patient's EHR in a location that will be accessible by the patient and ED provider. Each participating site will train patients and Emergency Department (ED) providers on how to access the IPP in the Electronic Health Record. The following required elements will be included in the EHR-embedded IPP:
  * Genotype
  * Individual pain plan-preferred analgesic agent, route, dose and dosing interval, last update time
  * Name and contact information for the SCD provider
  If the enrolled patient has a VOE visit at a nonparticipating ED, the patient will be able to access their IPP via the web or the patient portal app through their EHR. However, data will not be collected from these visits.

SUMMARY:
The overall purpose of this proposed study is to improve management of vaso-occlusive episodes (VOEs) in adult EDs. We aim to implement NHLBI recommendations for VOE treatment by embedding Individualized Pain Plans (IPPs) in the electronic health record (EHR). The EHR-embedded IPP will serve as a record of patients' SCD genotype and will include analgesic medication recommendations developed by the SCD provider. In this project, we will provide access to the IPP for both adult patients with SCD and ED providers. The proposed multisite study will use a pre-post study design, with a core set of mandatory intervention components and strategies for each participating site and optional components and strategies to allow for intervention adaptation to local needs and resources. The EHR-embedded IPP will be available for all adult ED providers to use as their routine practice, and patients will be invited to participate and enroll in the study. We will use a simplified Technology Acceptance Model to explain the use of the IPP and the RE-AIM framework to assess the Reach, Effectiveness, Adoption, Implementation, and Maintenance of the intervention.

DETAILED DESCRIPTION:
The study aims are as follows:

Aim 1: Assess the overall effectiveness of EHR-embedded IPPs on improving patient and provider outcomes associated with pain treatment in the adult ED setting. We will evaluate the effectiveness of the intervention on both patients and providers using a pre-post study design.

Sub-aim 1.a. To examine effectiveness of the EHR-embedded IPP on improving patients' perceived quality of ED pain treatment. We hypothesize that among enrolled patients with at least one ED VOE visit during the intervention period, the perceived quality of ED pain treatment will increase by 0.5 standard deviation (primary outcome) after an ED VOE visit when compared with the last ED VOE visits made by these patients within 90 days before enrollment. We will measure change pre- and post-intervention in secondary patient outcomes, including hospital admission rate within 12 months, ED VOE revisit rate, ED VOE readmission rate, and time to first dosage of pain medication provided in the ED.

Sub-aim 1.b. To examine the effectiveness of the EHR-embedded IPP on improving providers' self-efficacy in treating pain for patients with SCD and perceived quality of ED pain treatment. We hypothesize that the intervention will increase providers' self-efficacy in treating VOEs and managing pain for patients with SCD when compared with self-efficacy before the intervention. We will also explore the effect of the intervention on ED providers' perceived quality of ED pain treatment.

Aim 2: Assess the reach, adoption, implementation, and maintenance of the EHR-embedded IPP components and implementation strategies at each participating site. We will use the RE-AIM framework to evaluate intervention outcomes in addition to intervention effectiveness.

Sub-aim 2.a. To assess the reach of the EHR-embedded IPP. We will assess the reach of the intervention at the patient level by examining the proportion of patients enrolled in the study among all patients the team has reached out to recruit, and at the clinic level by examining the proportion of clinics participating in the intervention.

Sub-aim 2.b. To assess the adoption and implementation of the EHR-embedded IPP and track implementation strategies adopted by each site. We will assess the adoption of the intervention by examining characteristics of individual EDs that participate relative to the number of individual EDs affiliated with each study site who could have been recruited. We will assess implementation fidelity and outcomes, such as the proportion of eligible hematologists and nurse practitioners who receive IPP training, number of IPPs written and included in the EHR, required and optional intervention elements that are implemented as planned, IPP use by patients and providers, provider IPP adherence, and patients' and providers' perceived ease of use of the IPPs. We will track and report strategies used by participating sites through both quantitative data collection and qualitative interviews.

Sub-aim 2.c. To assess the intent to continue using the IPP from a multi-stakeholder perspective. We will assess patients' and providers' intent to continue using the IPP during the implementation period. At the end of the intervention, we will assess ED administrators' intent to continue using the IPP.

Aim 3: Assess organizational readiness at the beginning of the implementation and barriers and facilitators to the use of EHR-embedded IPPs. We will perform a Readiness Assessment to measure organization- and staff-level readiness at the beginning of the intervention to inform the selection and adaptation of implementation strategies. We will assess facilitators and barriers in adopting and implementing the IPPs from multiple stakeholder perspectives: patients, providers, and ED administrators.

Embedding IPPs in the EHR that are accessible to both ED providers and patients is a promising intervention to support the NHLBI evidence-based recommendations to guide treatment of VOE in the ED setting and improve quality of pain treatment in the ED and better patient outcomes. If EHR-embedded IPPs implemented and evaluated in this study show preliminary effectiveness, they could be scaled up within SCDIC Centers and expanded to other institutions outside the SCDIC. The results of this proposed study will accelerate the uptake of the NHLBI recommendation and establish standardized treatment in EDs for patients with SCD.

ELIGIBILITY:
Patient Inclusion Criteria:

* Age 18 years up to and including 45 years
* English speaking
* Confirmed SCD diagnoses . Confirmed is defined as supported by documentation in the medical record of a positive test for one of the following : Hb SS, Hb SC, Hb S -thalassemia, Hb SO, Hb SD, Hb SG, Hb SE, or Hb SF.
* Access to a cellular/mobile smart phone with access to text messaging (either Android or iPhone acceptable) .
* At least one Vaso-Occlusive Episode (VOE) visit to participating site Emergency Department (ED) the past 90 days from enrollment
* At least one visit at the study site sickle cell disease clinic within the past 12 months
* Willing and cognitively able to give informed consent

Patient Exclusion criteria:

* Patient's sickle cell provider states patient should not have a protocol or should not be administered opioids

Provider Inclusion Criteria:

* Provides pain treatment in one of the participating study Emergency Departments for a patient participant with a qualified ED visit .

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 279 (Actual)
Dates: Start 2020-10-27 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-10-01 (Actual)

PRIMARY OUTCOMES:
Change in Patient-perceived quality of ED pain treatment. | Baseline, 96 hours
  Three questions from the Adult Sickle Cell Quality of Life Measure (ASCQ-Me) and Quality of Care (QOC) measure will be used to measure the patient perceived quality of ED pain treatment

SECONDARY OUTCOMES:
ED revisit rate as measured by EHR retrieval | Day 7
ED revisit rate as measured by EHR retrieval | Day 30
Hospital readmission rate measured by EHR retrieval | Day 7
Hospital readmission rate measured by EHR retrieval | Day 30
Time to first dose of pain medication measured by EHR retrieval | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Paula Tanabe, PhD, Principal Investigator — Duke University School of Nursing
Locations (8):
- United States (8):
  - University of California San Francisco, Oakland, California
  - Georgia Regents University, Augusta, Georgia
  - University of Illinois, Chicago, Illinois
  - Washington University, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Duke University, Durham, North Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - St. Jude's, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: Yes
De-identified patient-level data will be available to researchers outside the SCDIC through an application and approval process as part of the SCDIC's Ancillary Studies Policy and Data Dissemination Plan. To protect the confidentiality and privacy of the participants, investigators granted access to the limited access data must adhere to strict requirements incorporated into a standard Data Use Agreement. In accordance with NHLBI policy, outside researchers will also be required to submit an approval tot RTI, the Data Coordinating Center, from their IRB.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available by RTI, the data coordinating center for the study, upon request.
Access Criteria: Researches outside of the SCDIC must submit requests for de-identified study related data to RTI, the data coordinating center.

REFERENCES:
- [Derived] Siewny L, King A, Melvin CL, Carpenter CR, Hankins JS, Colla JS, Preiss L, Luo L, Cox L, Treadwell M, Davila N, Masese RV, McCuskee S, Gollan SS, Tanabe P. Impact of an individualized pain plan to treat sickle cell disease vaso-occlusive episodes in the emergency department. Blood Adv. 2024 Oct 22;8(20):5330-5338. doi: 10.1182/bloodadvances.2023012439. PMID 38815230
- [Derived] Luo L, King AA, Carroll Y, Baumann AA, Brambilla D, Carpenter CR, Colla J, Gibson RW, Gollan S, Hall G, Klesges L, Kutlar A, Lyon M, Melvin CL, Norell S, Mueller M, Potter MB, Richesson R, Richardson LD, Ryan G, Siewny L, Treadwell M, Zun L, Armstrong-Brown J, Cox L, Tanabe P. Electronic Health Record-Embedded Individualized Pain Plans for Emergency Department Treatment of Vaso-occlusive Episodes in Adults With Sickle Cell Disease: Protocol for a Preimplementation and Postimplementation Study. JMIR Res Protoc. 2021 Apr 16;10(4):e24818. doi: 10.2196/24818. PMID 33861209